CLINICAL TRIAL: NCT03498833
Title: Comprehensive Knee Osteoarthritis Index (CKOAI): Scale Development, Validation and Reliability Testing
Acronym: CKOAI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maharishi Markendeswar University (Deemed to be University) (Other)
Responsible Party: Principal Investigator, Asir John Samuel, Associate Professor and Research Scholar, Maharishi Markendeswar University (Deemed to be University)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MMU/IEC/1021; U1111-1211-8513 (Other: Universal Trial Number); L-78484/2018 (Registry Identifier: Copyright Office (Government of India))
Record Dates: First submitted 2018-04-05; First posted 2018-04-17 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Osteo Arthritis Knee
Keywords: domains; item development; osteoarthritis; scale formulation; test retest reliability
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Intervention Model Description: All the domains and items in CKOAI will undergo reliability testing. Minimum 50 IKOA will be evaluated with the scale on two occasions within two weeks to establish test retest reliability. Cronbach's alpha for internal consistency and Intra class correlation coefficient for test retest reliability will be used to determine the degree of consistency of items in the scale. MDC will be calculated using the formulae, SEM = SD x √ (1-reliability) and MDC95 = √2 x (1.9) x (SEM). Significant level will be set at p value less than 0.05 (p < 0.05) to minimize the type-I error.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test-retest reliability testing (Other): Minimum 50 IKOA will be evaluated with the scale on two occasions within two weeks to establish test retest reliability.
  Interventions: Other: Test-retest reliability testing

INTERVENTIONS:
Other: Test-retest reliability testing — Set of patient reported outcome measures

SUMMARY:
Background:

Symptoms, balance, mobility, activities of daily life (ADL) and quality of life (QoL) are to be considered in rehabilitation of the individuals with knee osteoarthritis (IKOA). There are several scales to evaluate subjective perceptions and individual components in patients with osteoarthritis (OA). Till date, no scale is available to measure the combined balance, mobility, ADL and QoL in PKOA.

Objectives:

The objectives of the study are to develop a combined measure of symptoms, balance, mobility, ADL and QoL in PKOA, as comprehensive knee osteoarthritis index (CKOAI) and to validate the scale for its content, reliability and minimum detectable change (MDC)

Methods:

The study consists of a three stages. First stage is the scale (CKOI) item development and validation. This includes domain and item generating through systematic literature search to extract items related symptoms, balance, mobility, ADL and QoL in IKOA based on the International Classification of Functioning, Disability and Health (ICF) and through structured interviews. During scale validation, an expert panel will review the generated domains and items by Delphi Method, which will undergo revision and pilot testing. Based on the responsiveness of pilot testing will be revised finally. Second stage is to test re-test reliability. The third stage is to report the standard error of measurement (SEM) and minimal detectable change (MDC).

Data analysis:

All the domains and items in CKOAI will undergo reliability and criterion-related validity. Minimum 50 IKOA will be evaluated with the scale on two occasions within two weeks to establish test retest reliability. Cronbach's alpha for internal consistency and Intra class correlation coefficient for test retest reliability will be used to determine the degree of consistency of items in the scale. MDC will be calculated using the formulae, SEM = SD x √ (1-reliability) and MDC95 = √2 x (1.9) x (SEM). Significant level will be set at p value less than 0.05 (p < 0.05) to minimize the type-I error.

DETAILED DESCRIPTION:
Introduction:

One of the worldwide leading causes of disability and pain is osteoarthritis. 22% to 39% of 1.252 billion population suffer from osteoarthritis (OA). Hip and knee OA are the most prevalent forms of OA with the overall prevalence of knee OA is 28.7%. This will increase by 33.5% in 2030 due to alarming increase in aging population. Individuals with knee OA (IKOA) are seen with deficits in static and dynamic balance which comprises of impaired proprioception, muscle strength, disturbed postural control and decreased range of motion at knee joint. Furthermore, IKOA have pain and increase physical limitation and functional limitation. Eventually decreasing their quality of life (QoL).

Static balance in IKOA are assessed using several outcome measures such as, timed single-leg stance, functional reach test and variation of postural sway in unipedal or bipedal stance. More than two decade, Berg Balance Scale and Tinetti Performance-Oriented Mobility Assessment (balance subscale) were used to asses dynamic balance. Recently, Community Balance and Mobility Scale (CB&M) have been validated for the purpose. Isokinetic dynamometer has been in use for the purpose of estimating muscle strength. Proprioception was measured by joint repositioning test. Several researchers explored QoL in IKOA,and combined with functional independence.

Various measures of knee function adopted by International Knee Documentation Committee (IKDC) are subjective in nature. Patient reported problem based rating scale in IKOA with objective scoring is still lacking. There, the purpose of this research project is to develop a rating scale which does combine assessment of balance, mobility, ADL and QoL in IKOA.

Statement of the Problem:

The existing scales could not provide comprehensive assessment for balance, mobility, ADL and QoL in IKOA. Hence, there is a need to develop an objective scale to measure the above domains in IKOA

Purpose of the study:

The purpose of the study is to develop an objective combined assessment of symptoms, balance, mobility, ADL and QoL in IKOA (CKOAI) using systematic approach.

Objectives of the study:

1. To develop scale items and domains of CKOAI
2. To validate the developed scale for content validity
3. To estimate reliability of CKOAI
4. To report SEM and MDC

Procedure:

The study will be of cross-sectional observational study of scale validation. The study protocol was approved by the Institutional Ethics Committee of Maharishi Markandeshwar (Deemed-to-be) University (MMU/IEC/1021) on 8.12.2017. The study will consists of three major phases, comprising of item and domain generation, validation, reliability testing and estimating MDC.

Phase 1: Scale Development

Sub-Phase 1:Domain and item development:

1. Domain and item generating:

   using literature search and direct patient interviews.

   - Literature search: English language literature will be searched in databases.

   - Direct interview
2. Grouping item in domain Sub-phase 2: Content Validation

   * Using Delphi Method Sub-phase 3: First draft and scoring criteria Sub-phase 4: Pilot test Sub-phase 5: Revision Sub-phase 6: Final draft

Phase 2: Reliability testing

1. Check for internal consistency
2. Intra-rater reliability
3. Test-retest reliability

Phase 3: Estimating SEM and MDC

MDC will be calculated using the formulae, SEM = SD x √ (1-reliability) and MDC95 = √2 x (1.9) x (SEM). Significant level will be set at p≤ 0.05 to minimize the type-I error. For MCID, responsiveness of the scale will be determined on two occasions after regular conventional physiotherapy treatment of two week duration.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with osteoarthritic changes of grade 1 and greater on knee radiograph (Kellgren and Lawrence)
* Individuals with unilateral or bilateral knee osteoarthritis
* Both male and female
* Individuals who able to understand simple command
* Individuals who are willing to participate

Exclusion Criteria:

* History of hip and knee replacement surgery
* History of knee arthroscopic surgery within 6 months
* Any neurologic and musculoskeletal condition which affect their movement or balance
* Comorbidities such as cancer or cardiovascular disease

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2019-02-12 (Actual); Study Completion 2019-02-13 (Actual)

PRIMARY OUTCOMES:
Change in Comprehensive Knee Osteoarthritis Index | two occasions within two weeks to establish test retest reliability
  Set of patient reported outcome measures

CONTACTS AND LOCATIONS:
Overall Officials: Kanimozhi D Narkeesh, PhD, Study Director — Maharishi Markandeshwar Institute of physiotherapy and Rehabilitation
Locations (1):
- Maharishi Markandeshwar Institute of physiotherapy and Rehabilitation, Ambāla, Haryana, India

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers. We are planned to publish the results in journal.